CLINICAL TRIAL: NCT06270082
Title: A First-in-Human (FiH) Study of IK-595, an Oral Dual MEK/RAF Inhibitor, in Patients With RAS-or RAF-altered Advanced Solid Tumors
Brief Title: Study of IK-595 in RAS- or RAF-altered Advanced Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Limited resources and strategic priorities
Sponsor: Ikena Oncology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IK595-001
Record Dates: First submitted 2024-01-31; First posted 2024-02-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor, Adult; Colorectal Cancer; Pancreatic Cancer; Malignant Melanoma; Ras (Kras or Nras) Gene Mutation; BRAF Gene Mutation; CRAF Gene Mutation; Non-Small Cell Lung Carcinoma; Thyroid Carcinoma; Gliomas, Malignant
Keywords: IK-595; RAS-MAPK Pathway; MEK Inhibitor; MEK/RAF Inhibitor
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung; Thyroid Neoplasms; Glioma

STUDY DESIGN:
Intervention Model Description: Dose Escalation: BOIN design Dose Expansion: 4 genetically/molecularly defined cohorts using Simon 2-stage adaptive design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IK-595 (Experimental): Dose Escalation and Dose Expansion
  Interventions: Drug: IK-595

INTERVENTIONS:
Drug: IK-595 — Oral tablet administered in 28-day or 30-day cycles until treatment discontinuation criteria are met.

SUMMARY:
This is a Phase 1, FIH, Dose Escalation and Dose Expansion study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) effects, and preliminary antitumor activity of IK-595, a MEK/RAF molecular glue, administered orally as monotherapy in patients with advanced solid tumors with gene alterations in the RAS- MAPK pathway for whom there are no further treatment options known to confer clinical benefit.

DETAILED DESCRIPTION:
This is a Phase 1, FiH clinical study to evaluate the safety, tolerability, PK and pharmacodynamic effects, and preliminary anti-tumor activity of IK-595, a dual mitogen-activated protein kinase kinase (MEK)/ RAF kinase inhibitor, administered orally (PO) as monotherapy in patients with advanced solid tumors with gene alterations in the RAS- MAPK pathway for whom there are no further treatment options known to confer clinical benefit.

The study consists of an initial Dose Escalation phase using a Bayesian Optimal Interval (BOIN) design, followed by a Dose Expansion phase in 4 genetically/molecularly defined cohorts using 2-stage adaptive design.

During the Dose Escalation phase, backfilling may occur, where ≥ 3 additional patients can be enrolled at a given dose level once that dose level is deemed safe and tolerable by the Safety Review Committee. Backfilling includes, but is not limited to, patients with the following diagnoses: neuroblastoma RAS viral oncogene homolog-mutant (NRASmut) colorectal carcinoma (CRC), NRASmut malignant melanoma , Kirsten rat sarcoma viral oncogene homolog-mutant (KRASmut) CRC, KRASmut pancreatic cancer, KRASmut non-small cell lung cancer(NSCLC), B-Raf proto-oncogene, serine/threonine kinase-mutant (BRAFmut) Class II/III or BRAF fusion positive solid tumors, and Raf-1 proto-oncogene, serine/threonine kinase-mutant (CRAFmut) or fusion positive solid tumors.

Various dose levels and schedules will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age.
2. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
3. Adequate organ function as follows (specimens must be collected during the Screening Period within 7 days prior to entering the Treatment Period):

   1. ANC ≥ 1000/μL
   2. Hemoglobin > 9 g/dL
   3. Platelet count > 75,000/μL
   4. Calculated creatinine clearance ≥ 60 mL/min (using the Cockcroft-Gault formula or using other formulae per institutional guidelines)
   5. Serum total bilirubin ≤ 1.5 × ULN or direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 × ULN. Known Gilbert syndrome is allowed if total bilirubin is <3 × ULN
   6. AST and ALT ≤ 2.5 × ULN (or ≤ 5 × ULN if liver function abnormalities are due to underlying liver metastases)
   7. Coagulation: ≤ 1.5 × ULN unless patient is receiving anticoagulant therapy, as long as prothrombin time, international normalized ratio, or activated partial thromboplastin time is within therapeutic range of intended use of anticoagulants when applicable
4. Left ventricular ejection fraction ≥ 50% by echocardiogram or radionuclide test.
5. Patients must have recovered from the side effects of prior cancer-specific therapy to a minimum of ≥ Grade 1 by NCI-CTCAE version 5.0 criteria or return to baseline. Exceptionally, patients with ≤ Grade 2 neuropathy or other TRAEs may be eligible after discussion with the Sponsor.
6. Washout period since receipt of the last dose of prior anticancer therapy (including other investigational therapy):

   1. Checkpoint inhibitors such as cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), programmed cell death protein 1 (PD-1), or programmed death ligand 1 (PD-L1) inhibitors: ≥ 4 weeks
   2. For all other biologic agents (e.g., antiangiogenics): ≥ 3 weeks or a minimum of their dosing interval if shorter than 3 weeks (e.g., agents administered every 2 weeks would require a 2-week washout period)
   3. All other investigational agents: ≥ 4 weeks or ≥ 5 × t1/2, whichever is shorter.
7. If feasible, patients must be willing to consent to the submission of formalin-fixed paraffin-embedded (FFPE) tissue blocks of tumor tissue, preferably from a pretreatment, fresh tumor biopsy. Alternatively, archival tumor FFPE blocks or, ≥ 20 unstained slides of tumor tissue from available archival sources that are < 2 years old are acceptable.
8. Highly effective contraception for both male and female patients from Screening through 5 months after the last dose of study drug if the possibility of conception exists.
9. Patient or their legally acceptable representative must be able and willing to:

   1. Provide Institutional Review Board-or Institutional Ethics Committee-approved written informed consent in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal patient care.
   2. Comply with the study protocol and with the planned biopsy procedures.

   Inclusion Criteria for Dose Escalation Patients
10. Patients must have histologically or cytologically confirmed solid tumor malignancies that are advanced and unresectable, or metastatic with no available therapy known to confer clinical benefit, as evaluated by the treating physician. There is no upper limit on the number of prior lines of anticancer therapy received. Tumors must have confirmed RAS/RAF gene alterations as determined by next-generation sequencing or fluorescence in situ hybridization, as documented by local testing:

    1. NRASmut solid tumors, including but not limited to melanoma, CRC, and others
    2. KRASmut solid tumors, including but not limited to NSCLC, pancreatic carcinoma, and CRC
    3. BRAFmut Class I/II/ III or BRAF fusions solid tumors, including but not limited to melanoma, NSCLC, thyroid carcinoma
    4. CRAF-altered solid tumors (mutations and gene fusions)
    5. NF1mut solid tumors, including but not limited to nerve sheath tumors, gliomas, malignant melanoma, breast cancer, and others
11. Patients who have measurable or evaluable disease by RECIST 1.1 criteria, as assessed by the Investigator/local radiologist.

    Inclusion Criteria for Dose Expansion Patients
12. All patients must have a histological diagnosis of an advanced, unresectable, locally recurrent, or metastatic disease with no available therapy known to confer clinical benefit, as evaluated by the treating physician. There is no upper limit on the number of prior lines of anticancer therapy received.
13. Patients must be enrolled in 1 of the following 4 dose expansion cohorts:

    1. Cohort 1: Molecularly confirmed NRASmut CRC as determined by local test results
    2. Cohort 2: Molecularly confirmed NRASmut malignant melanoma as determined by local test results
    3. Cohort 3 Molecularly confirmed KRASmut NSCLC as determined by local test results
    4. Cohort 4: Any solid tumors with molecularly confirmed pathogenic BRAF non-V600X mutations or fusions, or pathogenic CRAF mutations or fusions as determined by local test results
14. Patients must have ≥ 1 measurable lesion per RECIST 1.1 criteria as assessed by the Investigator/local radiologist. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions. Exceptionally, patients with tumors that are evaluable but non-measurable per RECIST 1.1 criteria can be enrolled following approval by the Sponsor.

Exclusion Criteria:

1. Patients with any active central nervous system (CNS) lesion either symptomatic or radiologically unstable and/or leptomeningeal metastasis. However, patients previously treated for these conditions that have had stable CNS disease (verified with consecutive imaging studies) for > 3 months, are asymptomatic and are not currently taking corticosteroids, or are on stable dose or decreasing of corticosteroids for ≥ 7 days prior to enrollment are eligible.
2. Patients who have not recovered to ≤ Grade 1 or baseline from all AEs due to prior anticancer therapies. Exceptionally, patients with ≤ Grade 2 neuropathy or other TRAEs may be eligible after discussion with the Sponsor.
3. Any other concurrent antineoplastic treatment or investigational agent except for localized radiation therapy for symptom palliation (to be considered nontarget lesions after treatment) and/or hormonal therapy for ductal DCIS/LCIS/Stage 1 breast cancer that has been stable on therapy for ≥ 3 years.
4. Uncontrolled or life-threatening symptomatic concomitant disease (including known symptomatic HIV-positive with an active AIDS-defining opportunistic infection or a current CD4 count < 350 cells/μL; symptomatic active hepatitis B or C checked at screening; or active tuberculosis). Patients with HIV are eligible if:

   1. They have received antiretroviral therapy (ART) as clinically indicated for ≥ 4 weeks prior to entering the Treatment Period of the study;
   2. They continue on ART as clinically indicated while on study;
   3. CD4 counts and viral loads are monitored per standard of care by a local health care provider.
5. Has received prior radiotherapy for palliation ≤ 2 weeks prior to the first dose of study treatment. Patients must have recovered from all radiation-related toxicities.
6. History of a second malignancy requiring systemic treatment ≤ 3 years prior to enrollment. Patients who have remained cancer-free ≤ 3 years of enrollment are eligible. Patients with history of prior early stage basal/squamous cell skin cancer or noninvasive or in situ cancers that have undergone definitive treatment at any prior time are eligible.
7. Clinically significant cardiovascular disease:

   1. Cerebral vascular accident/stroke (< 6 months prior to enrollment)
   2. Myocardial infarction (< 6 months prior to enrollment)
   3. Unstable angina (< 6 months prior to enrollment)
   4. Congestive heart failure (New York Heart Association Classification Class III or IV)
   5. The presence of any condition that can increase proarrhythmic risk (e.g., hypokalemia, bradycardia, heart block), including any new, unstable, or serious cardiac arrhythmia requiring medication, or other baseline arrhythmias that might interfere with interpretation of ECGs on study (e.g., bundle branch block).
   6. Patients with QT interval corrected by Fridericia's formula (QTcF) > 470 msec for both men and women on screening ECG are excluded. Patients with a bundle branch block must have QT interval corrected for bundle branch block.
   7. Patients who are on stable doses of concomitant medication with known prolongation of QTcF if QTcF is > 470 msec.
8. Known previous or current serious ophthalmic disorders, including history of glaucoma, history of retinal vein occlusion (RVO) or current risk factors for RVO, history of retinal pathology or evidence of retinal pathology.
9. Active skin disorder requiring systemic treatment ≤3 months prior to start of study treatment.
10. History of rhabdomyolysis ≤3 months prior to start of study treatment.
11. Patients taking any medication on the prohibited medication list are excluded from the study unless they can be transferred to other medications.
12. Has an active infection requiring systemic therapy.
13. A woman of childbearing potential who has a positive pregnancy test prior to initiating study treatment.
14. Breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the Screening visit through 5 months after the last dose of study treatment.
15. Patients who are unable to swallow or retain oral medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events, including treatment-related adverse events, and serious adverse events | From treatment initiation through study completion, average of 36 months
  • Frequency and severity of treatment-emergent adverse events, including treatment-related adverse events, and serious adverse events
Dose Limiting Toxicities | The first 30 days of treatment for each patient during Dose Escalation
  Number of patients with dose-limiting toxicities (Dose Escalation only)
Treatment-Emergent Adverse Events | From treatment initiation through study completion, average of 36 months
  Number and percentage of patients with ≥ 1 treatment-emergent adverse events leading to dose modifications and treatment discontinuation
Recommended Phase 2 Dose (RP2D) and/or maximum tolerated dose (MTD) of IK-595 | From treatment initiation through dose escalation, approximately 1 year
  Selection of dose level to take proceed with in Dose Expansion and/or Phase 2

SECONDARY OUTCOMES:
Pharmacokinetics of IK-595: half-life (t1/2) | From treatment initiation through dose escalation, approximately 1 year
  half-life (t1/2)
Pharmacokinetics of IK-595: Area Under the Curve (AUC) | Approximately 1 year
  AUC
Pharmacokinetics of IK-595: Maximum Plasma Concentration (Cmax) | Approximately 1 year
  Cmax
Pharmacokinetics of IK-595: Minimum Plasma Concentration (Cmin) | Approximately 1 year
  Cmin
To evaluate pERK fold change from baseline in paired tumor biopsies | Through study completion, average of 36 months
  To evaluate the pharmacodynamic effects of IK-595 on the levels of phosphorylated extracellular signal-regulated kinase (pERK) in paired tumor biopsies
Antitumor activity per RECIST 1.1: Disease control rate (DCR) of IK-595 as a single agent | Through study completion, average of 36 months
  Complete Response [CR] + Partial Response [PR] + stable disease ≥ 16 weeks
Antitumor activity per RECIST 1.1: Time to response (TTR) of IK-595 as a single agent | Through study completion, average of 36 months
  TTR
Antitumor activity per RECIST 1.1: Duration of response (DOR) of IK-595 as a single agent | Through study completion, average of 36 months
  DOR
Antitumor activity per RECIST 1.1: Objective response rate (ORR) of IK-595 as a single agent | Through study completion, average of 36 months
  ORR
Antitumor activity: Median progression-free survival (PFS) of IK-595 as a single agent | Through study completion, average of 36 months
  PFS

OTHER OUTCOMES:
Antitumor activity: Median overall survival (OS) of IK-595 as a single agent | Through study completion, average of 36 months
  OS

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Germa, MD, Study Chair — Ikena Oncology
Locations (15):
- United States (15):
  - City of Hope, Duarte, California
  - University of California Irvine, Orange, California
  - Sarah Cannon Research Institute at HealthOne, Denver, Colorado
  - Johns Hopkins University of Medicine Sidney Kimmel Comprehensive Care Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - START Midwest, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center- Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Next Oncology, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Next Oncology- San Antonio, San Antonio, Texas
  - INOVA Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No